CLINICAL TRIAL: NCT06651801
Title: A Pilot Randomized Controlled Trial Assessing the Feasibility and Acceptability of Group Medical Visits for Anxiety and Depression
Brief Title: Feasibility and Acceptability of Group Medical Visits for Anxiety and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Kirsten Penner-Goeke, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS26533
Record Dates: First submitted 2024-10-07; First posted 2024-10-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Mental Health Care; Anxiety and Depression; Pilot Study
Keywords: Group Medical Visits; Anxiety; Depression; Shared Medical Appointments; Pilot Study
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard client services (No Intervention): Participants will follow-up with their primary care provider (family physician or nurse practitioner).
- Virtual outpatient care (Experimental)
  Interventions: Behavioral: Group Medical Visits

INTERVENTIONS:
Behavioral: Group Medical Visits — Group medical visits occur every 2 weeks virtually (via Zoom) for 6 months. Each group consists of 45 minutes of group time and 5 minute individual check-in appointments. The group time consists of psychoeducation, group support, and medication follow-up.
  Arms: Virtual outpatient care

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and acceptability of the intervention, Group Medical Visits (GMVs), for patients with depression and anxiety. It also aims to get some initial information on the effectiveness of GMVs on reducing depression and anxiety scores, which will help inform power calculations for a future larger randomized controlled trial (RCT). The main question it aims to answer is:

* Are GMVs feasible and acceptable to patients with depression and anxiety?

This study consists of a pilot RCT with an intervention and control arm. At enrollment, participants will be randomized to the intervention group, 6 months of GMVs, or to the control group, which consists of "standard client services". For the GMV group, participants will engage in a biweekly virtual group that is similar to a standard psychiatric follow-up. Participants in the control group will receive standard care after a psychiatric assessment, which includes follow-up with their primary care provider (family physician or nurse practitioner), individual psychiatric care if suggested by the psychiatrist who did their psychiatric assessment, and/or a referral to publicly funded therapy groups if interested.

ELIGIBILITY:
Inclusion Criteria:

* Adult Central Intake patients (patients referred for psychiatric consultation by their primary care provider) whose primary mental health issue is an anxiety disorder (social anxiety, generalized anxiety, or panic disorder) or depression (major depressive disorder or persistent depressive disorder)
* Able to participate in English language group with up to 10 participants
* Able to commit to a virtual biweekly group for about 1.5 hours each group
* Able to do virtual group from a private location with camera access
* Live in community in Manitoba and plan to stay for 6-month period

Exclusion Criteria:

* Patients with Bipolar 1 or 2 Disorder (even if current episode depression)
* Primary diagnosis of a personality disorder leading to anxiety/depression symptoms (personality disorder traits are not an exclusion criteria)
* Patients who already have established longitudinal care with a psychiatrist
* Received ECT treatment within past 6 months
* Any diagnosis that would significantly impact ability to participate in the group. For example:
* Moderate-to-severe substance use disorders (in particular substance use throughout day or inability to attend group without using substances before)
* Current psychotic symptoms
* Moderate-to-severe intellectual disability or neurocognitive disorder
* Current significant eating disorder symptoms (for example resulting in significant weight loss/malnutrition or that take up a significant part of the day either mentally or physically)
* Self harm behaviour requiring medical/psychiatric attention or active suicidal ideation/suicide attempts within the past 6 months
* Concern about safety of other group members/facilitators if this patient were to join

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-4 Scale (CSQ-4) | Month 3 and month 6 of intervention
  Includes 4 items that measure client satisfaction. Items are rated on a 4-point scale, with total score ranging from 4 to 16. A higher score indicates higher satisfaction.
Recruitment and Retention Rate | Baseline, during the intervention, through study completion (estimation 9 months)
  The investigators will examine the rates of how many participants sign up and are enrolled in the program, along with the drop-out rate throughout the program.
Primary Care Provider Satisfaction with Psychiatric Care | Month 6 of intervention
  The investigators will conduct a telephone survey with the primary care providers (PCPs) of the participants who were randomized to the intervention group. The survey will assess how satisfied the PCPs are with the care that their patient received during the trial. The survey consists of one question assessing overall satisfaction, rated on a 5-item scale from "Very Satisfied" to "Very Dissatisfied", two open ended questions assessing which aspects of care the PCPs were satisfied and not satisfied with, and 5 questions assessing whether they would refer other patients to the program, what benefits were there of having their patient in the program, and what aspects of the program could be improved.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Enrolment (before randomization), baseline (before intervention), month 3, and month 6 of intervention
  Includes 9 items assessing depressive symptom severity. Total score ranges from 0 to 20, with a higher score indicating higher symptom severity.
General Anxiety Disorder-7 (GAD-7) | Enrolment (before randomization), baseline (before intervention), month 3, and month 6 of intervention
  Includes 7 items assessing anxiety symptom severity. Total score ranges from 0 to 21, with a higher score indicating higher symptom severity.
Recovery Assessment Scale 24 (RAS24) | Enrolment (before randomization), baseline (before intervention), month 3, and month 6 of intervention
  Includes 24 items assessing personal recovery. Total score ranges from 24 to 120, with higher scores indicating higher levels of recovery.
Mental Health Quality of Life Questionnaire (MHQoL) | Enrolment (before randomization), baseline (before intervention), month 3, and month 6 of intervention
  Consists of 7 domains with 4 items assessing each. Total score ranges from 0 to 21, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- PsycHealth Centre, Winnipeg, Manitoba, Canada